CLINICAL TRIAL: NCT05287087
Title: My Symptoms - Feasibility Study: Feasibility of Intervention and Evaluation of an eHealth and GP Assisted Programme for Persistent Symptoms in Primary Care for Persistent Symptoms in Primary Care
Brief Title: My Symptoms - Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Rosendal, Senior researcher, PhD, General Practitioner, Aarhus University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1-10-72-372-21
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Persistent Physical Symptoms
MeSH Terms: interventions — E1A-Associated p300 Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: We will inform GPs about the possibility of being assigned to one of two interventions expected to have each their advantages and disadvantages, hence being of equal value to patients. The GPs will know the content of their assignment but will not be informed about the specific content of the other intervention. Enrolled patients will only be informed whether they are to use the programme My Symptoms 1 or My Symptoms 2 accessed via a website.
  Outcome assessment and data analyses in this feasibility study conducted by the project researchers will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Symptoms 1 (MySt-1) (Active Comparator): GPs will receive an introduction to the overall content of the eHealth programme MySt-1. The information will be given to participating GPs and their staff during a 1½-hour session in the practice. The research assistant will go through the logistics of the patient recruitment and evaluation step-by-step and GPs and relevant staff will subsequently have access to the programme.
  The patients will get access to a basic eHealth programme (My Symptoms 1). The programme is an internet-delivered self-help programme supporting patients' selfefficacy and behavioural changes. The programme is activated by the patient after prescription by the GP.
  Interventions: Behavioral: My Symptoms 1 (MySt-1)
- My Symptoms 2 (MySt-2) (Experimental): GPs will attend a one-day training course of 7 hours including: in depth insight into the My Symptoms 2 eHealth programme, comprehensive understanding of PPS, training of communication skills and the use of contextual (non-specific/common psychological) factors. The training programme has been developed in cooperation with the national GP association offering CME (PLO-e). Lecturers and trainers will be GPs and psychologists from the research team.
  The patients will get access to an advanced eHealth programme (My Symptoms 2). The programme is an internet-delivered self-help programme supporting patients' selfefficacy and behavioural changes. The programme is activated by the patient after prescription by the GP.
  Interventions: Behavioral: My Symptoms 2 (MySt-2)

INTERVENTIONS:
Behavioral: My Symptoms 1 (MySt-1) — The patients will get access to an eHealth programme consisting of:
  1. A questionnaire including the BDS checklist
  2. A brief introductory animation about how to understand symptoms in general
  3. Basic information on symptom in general and on six common symptoms: headache, fatigue, dizziness, pain, dyspepsia and abdominal unease.
  4. A brief animation about the interaction of body and mind.
  These four provisions are identical to the first part of the MySt-2.
  Arms: My Symptoms 1 (MySt-1)
Behavioral: My Symptoms 2 (MySt-2) — The patients will get access to an eHealth programme consisting of:
  1. A questionnaire including the BDS checklist
  2. A brief introductory animation about how to understand symptoms in general
  3. Basic information on symptom in general and on six common symptoms: headache, fatigue, dizziness, pain, dyspepsia and abdominal unease.
  4. A brief animation about the interaction of body and mind.
  5. Thorough symptom explanations
  6. Physical energy (focus on sleep, diet and activity)
  7. Values and choices (focus on meaning and existential issues)
  8. Emotional health (focus on emotion regulation)
  9. Mental energy (focus on stress regulation and thinking)
  After 4-6 weeks, the patient will see the GP for a follow-up consultation.
  Arms: My Symptoms 2 (MySt-2)

SUMMARY:
The proposed project 'My Symptoms' is part of a large research programme: eHealth and GP-assisted self-help interventions for persistent physical symptoms (eASY). See www.minesymptomer.dk.

The research programme is an ambitious and dedicated effort aiming at improvement of functioning and quality of life for individuals with persistent physical symptoms (PPS) and prevention of the development of chronic functional disorders and associated loss of working capacity and high use of health care. At present, access to specialized treatment of PPS is very limited and treatment capacity in general practice is restricted to brief consultations - often with poor opportunity to make a treatment plan for symptoms. In order to improve health care for patients with PPS, the investigators have developed a web-based selfhelp programme for symptoms. As part of the intervention, this programme is prescribed by the patient's general practitioner (GP). The investigators have applied a high degree of user involvement (GPs and patients) in the development process but there is a need to evaluate how the new treatment programme is in fact adopted and how it affects GPs in routine care and patients in daily life. With this study, the investigators wish to take the first step towards a comprehensive and rigorous evaluation. Results from this feasibility study will both qualify a subsequent randomised controlled trial (RCT) in a larger pilot study and provide information for a potential national dissemination.

DETAILED DESCRIPTION:
Drawing on existing evidence about symptoms, functional disorders and eHealth interventions combined with user involvement, the investigators have developed a web-based self-help programme for PPS: "My Symptoms". The programme builds on the bio-psycho-socialexistential illness model and enhanced cognitive behavioural theory. Seven treatment modules focus on psychoeducation, lifestyle intervention, self-regulation and graded exercise delivered through text, videos, animations and audio files (see overview of content in table 1). Furthermore, it includes a 1-day course for GPs and a mandatory follow-up appointment between patient and GP at the programme closure. The training course for the GPs will focus on patient identification, positive reinforcement and familiarity with the content of the programme. The programme must be prescribed by GPs and is recommended to use for 6 weeks.

The objectives with the present feasibility study are: 1) to test and refine the GP training course, 2) to explore the planned logistics for patient recruitment, 3) to evaluate GP and patient questionnaires, and 4) to evaluate patients' use of the programme and 5) follow-up consultations with their GP.

With regard to 2-5, the following questions will be adressed and explored:

1. Which modifications are needed to the predefined procedures for consecutive patient enrolment?
2. What are the results of patient enrolment with respect to recruitment rates and patient characteristics? (Patients are asked and screened consecutively, but how many accept participation and fulfil inclusion criteria? What characterises enrolled patients compared to refusers?)
3. To what extent do patients accept and engage with the baseline research questionnaires?
4. When do included patients engage with the programme after enrolment (delay in time)?
5. How much do included patients interact with the intervention, i.e. how many patients log into the program, which modules and pages are accessed, and how many tools are used?
6. How many patients consult the GP for a follow-up consultation and when does this consultation take place?
7. How many contacts do the patients have to participating practices during their use of the programme?

Alongside this part of the feasibility study, the investigators will conduct a separate in-depth qualitative study (field study observations and interviews) on GP and patient interactions with the intervention. A separate protocol has been developed for this part of the feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Listed with participating practice
* Giving informed consent to participation in the study
* Consulting a GP or GP supervised staff
* Multiple symptoms, i.e. 4 or more symptoms within the past 4 weeks, according to the Bodily Distress Syndrome checklist (a validated symptom checklist with 25 items)

Exclusion Criteria:

* Not consulting for symptoms
* Symptoms are due to acute disease
* Symptoms must primarily be treated by medicine or surgery
* Not eligible due to language or cognitive problems
* Patient severely affected by other disease
* Other, GP assessment/statement (e.g.: All symptoms are with recent onset and I see no need for intervention at present, I do not believe the patient will benefit the least bit from participation in the eHealth programme at this time)
* Patient declines to use the eHealth program despite GP recommendation
* Patient has not accessed the programme within 2 weeks from referral from the GP

Criteria for stratification:

- Long-term sick leave, i.e. more than 8 weeks, will be a criterion for stratification in order to enable analyses on the target group of patients with PPS without chronicity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients in the target age group visiting the practice | Recruitment (Week 1)
Number of patients refusing participation | Recruitment (Week 1)
Number of patients fulfilling the inclusion criteria | Recruitment (Week 1)
Number of patients excluded by the GPs and reasons for this | Recruitment and/or referral consultation (Week 1-3 expectedly)
Number of patients not accepting the invitation for intervention despite consent to participate in the project (drop-outs) | Invitation for referral consultation/at referral consultation (Week 1-3 expectedly)
Number of patients who do not log into the programme within 2 weeks from referral or only log into the programme once (drop-outs) | 2 weeks after referral consultation (Week 4-5 expectedly)

SECONDARY OUTCOMES:
Symptoms | Recruitment (screening), programme login (baseline), end of treatment
  Bodily Distress Syndrome checklist
Symptom intensity and interference | Recruitment (screening), programme login (baseline), end of treatment
Illness perception | Recruitment (screening), programme login (baseline), end of treatment
  Illness Perception Questionnaire
Anxiety and Depression | Recruitment (screening), programme login (baseline), end of treatment
  Symptom Checklist (SCL)-13
Health anxiety | Recruitment (screening), programme login (baseline), end of treatment
  Whiteley-6R
Global health | Recruitment (screening), programme login (baseline), end of treatment
  One item from SF-36
Evaluation of GP at referral consultation | Programme login (baseline)
  6 items
Program expectations | Programme login (baseline)
  2 items adapted from the Credibility Expectancy Questionnaire
Quality of life | Programme login (baseline), end of treatment
  SF-36
Quality of life | Programme login (baseline), end of treatment
  EQ-5D-5L (EuroQol)
Pain self-efficacy | Programme login (baseline), end of treatment
  Pain Self-Efficacy Questionnaire
Illness behavior | Programme login (baseline), end of treatment
  The Behavioural Responses to Illness Questionnaire
Productivity Costs | Programme login (baseline), end of treatment
  Productivity Costs Questionnaire (IMTA)
Health care utilization | Programme login (baseline), end of treatment
  Medical Consumption Questionnaire (IMTA)
Program evaluation | End of treatment
  13 items
Global impression of change | End of treatment
  1 item
Evaluation of GP at referral consultation | End of treatment
  2 items

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Program access for patients — https://mine-symptomer.dk/